CLINICAL TRIAL: NCT04259749
Title: Experimentally Testing Legally Feasible Regulatory Options for Reducing the Impact of the Point-of-sale Retail Environment on Adolescent Tobacco Use
Brief Title: Testing Legally Feasible Options: Study 1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RAND (Other)
Responsible Party: Principal Investigator, William Shadel, Senior Behavioral Scientist, RAND
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R01CA236608 (NIH)
Record Dates: First submitted 2020-02-02; First posted 2020-02-06 (Actual); Results first posted 2023-10-30 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Tobacco Use
MeSH Terms: conditions — Tobacco Use

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Status Quo (Active Comparator): The StoreLab power wall will display all tobacco products.
  Interventions: Other: All flavored and mentholated products available
- Flavors Banned (Experimental): The StoreLab will display tobacco products without characterizing flavors, but will allow mint and menthol products to be displayed.
  Interventions: Other: Flavor Ban
- Flavors and Menthol Banned (Experimental): The StoreLab will display only tobacco products without characterizing flavors; mint and menthol will not be displayed.
  Interventions: Other: Flavor Ban; Other: Menthol Ban

INTERVENTIONS:
Other: Flavor Ban — Only flavored tobacco products are banned
  Arms: Flavors Banned; Flavors and Menthol Banned
Other: Menthol Ban — Mentholated products are banned
  Arms: Flavors and Menthol Banned
Other: All flavored and mentholated products available — No bans: All tobacco products are available
  Arms: Status Quo

SUMMARY:
The overall aim of this research is to experimentally evaluate different, legally-viable approaches to reducing the impact of the point-of-sale (POS) retail environment on adolescent tobacco use risk. This study will be investigating the regulations for four classes of tobacco products (cigarettes, e-cigarettes, smokeless tobacco, little cigars/cigarillos). Study 1 (study 1 out of 3 proposed) will examine whether eliminating the sale of flavored tobacco products at POS reduced adolescents' tobacco use risk.

DETAILED DESCRIPTION:
Tobacco advertising at retail point-of-sale (POS) includes promotional allowances that permit tobacco products to be advertised and sold at reduced cost to consumers (e.g., two-for-one specials); high visibility sale and therefore placement of hundreds of tobacco products on power walls; and the display of a large, diverse collection of poster advertisements on the exterior of the stores. Adolescents are at significant risk for having repeated exposures to this tobacco rich POS environment and such exposures contribute to increases in adolescent tobacco use. Although curbing the effect of the tobacco rich POS environment on adolescent tobacco use is a critical public health goal, some POS advertising regulations are unlikely to be viable in the United States because they impinge upon the tobacco industry's commercial free speech rights. For example, eliminating the tobacco power wall is probably not a viable option in the US as it has been successfully challenged in court by the tobacco industry. POS regulations that do not violate the industry's commercial free speech rights stand a better chance of being upheld by the courts. For example, eliminating tobacco product price promotions, reducing the availability of tobacco products by restricting the sale of flavored products, and restricting how much door/window space tobacco product posters can occupy at POS, all have been implemented as feasible and legally defensible regulatory options at POS. The evidence base supporting the efficacy of these initiatives is, however, almost non-existent - leaving them open to legal scrutiny. The overall aim of this research is to experimentally evaluate different, legally-viable approaches to reducing the impact of the POS retail environment on adolescent tobacco use risk. This research will be investigating the regulations for four classes of tobacco products (cigarettes, e-cigarettes, smokeless tobacco, little cigars/cigarillos): the extent to which eliminating tobacco product price promotions (Study 2), restricting how much door/window space tobacco posters can occupy at POS (Study 3), and eliminating the sale of flavored and/or mentholated tobacco products (Study 1) reduce adolescent tobacco-use risk. Each study will evaluate for possible gender and race (African-American vs Caucasian) differences. The studies will take place in the RAND StoreLab, a life-sized replica of a convenience store that was developed to experimentally evaluate how altering aspects of tobacco promotion at POS influences tobacco use. The present record is for Study 1.

ELIGIBILITY:
Inclusion Criteria:

* ages 11-20, parental consent/adolescent assent for minors

Exclusion Criteria:

* any medical or psychiatric condition which would make compliance with the study protocol difficult (based on parent report).
* Previous participation (by either adolescent or parent) in a previous StoreLab study

Ages: 11 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 267 (Actual)
Dates: Start 2020-01-16 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William G Shadel, PhD, Principal Investigator — RAND
Locations (1):
- RAND, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Status Quo | Flavors Banned | Flavors and Menthol Banned
Started | 89 | 91 | 87
Completed | 89 | 91 | 87
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Status Quo | Flavors Banned | Flavors and Menthol Banned | Total
Number analyzed (Participants) | 89 | 91 | 87 | 267
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.73 (3.23) | 16.47 (3.26) | 16.56 (3.11) | 16.56 (3.11)
Sex/Gender, Customized [Number; unit: participants]
  male | 24 | 28 | 31 | 83
  female | 61 | 62 | 51 | 174
  other/nonbinary | 4 | 1 | 5 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 4 | 6 | 16
  Not Hispanic or Latino | 83 | 86 | 81 | 250
  Unknown or Not Reported | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 13 | 18 | 13 | 44
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 7 | 7 | 18 | 32
  White | 59 | 54 | 52 | 165
  More than one race | 7 | 9 | 3 | 19
  Unknown or Not Reported | 3 | 3 | 1 | 7
Region of Enrollment [Number; unit: participants]
  United States | 89 | 91 | 87 | 267

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants Susceptible to Smoking Cigarettes After Shopping in the StoreLab (Non-flavored)
Description: Self-report items: "Do you think you will try an unflavored cigarette (unflavored = cigarettes without menthol or mint) anytime soon?", "Do you think you will smoke an unflavored cigarette (unflavored = cigarettes without menthol or mint) anytime in the next year?"; and "If one of your best friends offered you an unflavored cigarette (unflavored = cigarettes without menthol or mint), would you smoke it?". Responses to each item are made on a 1 (Definitely Not) to 10 (Definitely Yes) scale and the three items were summed for a total scale score. The total scale score was dichotomized: those who scored a '3' were recoded as '0' (not susceptible) and any scores greater than '3' were coded as '1' (susceptible). Proportion of susceptible participants was the outcome (number susceptible over the total number of participants within condition).
Time Frame: There is one visit in this research: This variable is assessed at that visit, immediately after the experimental manipulation.
Population: The numbers of participants per condition differs from the baseline table because of missing data.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Status Quo | Flavors Banned | Flavors and Menthol Banned
Number analyzed (Participants) | 74 | 73 | 74
proportion of participants | .18 [.10 to .30] | .23 [.14 to .36] | .33 [.21 to .48]
Statistical Analysis 1: Comparison: Status Quo vs Flavors Banned; Test type: Other; Odds Ratio (OR) = 1.40, 95% CI 2-sided [0.58 to 3.40] — Adjusted for age, education, lifetime use of tobacco products
Statistical Analysis 2: Comparison: Status Quo vs Flavors and Menthol Banned; Test type: Other; Odds Ratio (OR) = 2.28, 95% CI 2-sided [0.92 to 5.63] — Adjusted for age, education, and lifetime use of tobacco products

2. Primary Outcome: Proportion of Participants Susceptible to Smoking Cigarettes After Shopping in the StoreLab (Menthol)
Description: Self-report items: "Do you think you will try a cigarette flavored with menthol or mint anytime soon?", "Do you think you will smoke a cigarette flavored with menthol or mint anytime in the next year?"; and "If one of your best friends offered you a cigarette flavored with menthol or mint, would you smoke it?". Responses to each item were made on a 1 (Definitely Not) to 10 (Definitely Yes) scale and the three items were summed. The total scale score was dichotomized: those who scored a '3' were recoded as '0' (not susceptible) and any scores greater than '3' were coded as '1' (susceptible). Proportion of susceptible participants was the outcome (number susceptible over the total number of participants within condition).
Time Frame: as for outcome 1
Population: The numbers of participants per condition differs from the baseline table because of missing data.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Status Quo | Flavors Banned | Flavors and Menthol Banned
Number analyzed (Participants) | 75 | 72 | 76
proportion of participants | .13 [.06 to .23] | .19 [.10 to .32] | .33 [.21 to .48]
Statistical Analysis 1: Comparison: Status Quo vs Flavors Banned; Test type: Other; Odds Ratio (OR) = 1.58, 95% CI 2-sided [0.61 to 4.07] — Adjusted for age, education, and lifetime use of tobacco products
Statistical Analysis 2: Comparison: Status Quo vs Flavors and Menthol Banned; Test type: Other; Odds Ratio (OR) = 3.45, 95% CI 2-sided [1.32 to 9.02] — Adjusted for age, education, and lifetime use of tobacco products

3. Secondary Outcome: Proportion of Participants Susceptible to Using Electronic Nicotine Delivery Device (ENDS) After Shopping in the StoreLab (Non-flavored)
Description: Self-report items: "Do you think you will try an unflavored vaping product soon?", "Do you think you will use an unflavored vaping product anytime in the next year?"; and "If one of your best friends offered you an unflavored vaping product would you use it?". Responses to each item were made on a 1 (Definitely Not) to 10 (Definitely Yes) scale and the three items were summed. The total scale score was dichotomized: those who scored a '3' were recoded as '0' (not susceptible) and any scores greater than '3' were coded as '1' (susceptible). Outcome is number of participants susceptible to using ENDS after shopping in the StoreLab (non-flavored). Proportion of susceptible participants was the outcome (number susceptible over the total number of participants within condition).
Time Frame: as for outcome 1
Population: The numbers of participants per condition differs from the baseline table because of missing data.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Status Quo | Flavors Banned | Flavors and Menthol Banned
Number analyzed (Participants) | 74 | 71 | 75
proportion of participants | .17 [.09 to .28] | .23 [.13 to .36] | .34 [.22 to .49]
Statistical Analysis 1: Comparison: Status Quo vs Flavors Banned; Test type: Other; Odds Ratio (OR) = 1.48, 95% CI 2-sided [.59 to 3.68] — Adjusted for age, education, and lifetime use of tobacco
Statistical Analysis 2: Comparison: Status Quo vs Flavors and Menthol Banned; Test type: Other; Odds Ratio (OR) = 2.60, 95% CI 2-sided [1.05 to 6.42] — Adjusted for age, education, and lifetime use of tobacco products

4. Secondary Outcome: Proportion of Participants Susceptible to Using Electronic Nicotine Delivery Device (ENDS) After Shopping in the StoreLab (Sweet-flavored)
Description: Self-report items: "Do you think you will try a vaping product flavored with fruit, candy, alcohol or non-alcohol drink, or some other sweet flavor soon?", "Do you think you will use a vaping product flavored with fruit, candy, alcohol or non-alcohol drink, or some other sweet flavor anytime in the next year?"; and "If one of your best friends offered you a vaping product flavored with fruit, candy, alcohol or non-alcohol drink, or some other sweet flavor, would you use it?". Responses to each item were made on a 1 (Definitely Not) to 10 (Definitely Yes) scale and the three items were summed. The total scaled score was dichotomized: those who scored a '3' were recoded as '0' (not susceptible) and any scores greater than '3' were coded as '1' (susceptible). Proportion of susceptible participants was the outcome (number susceptible over the total number of participants within condition).
Time Frame: as for outcome 1
Population: The numbers of participants per condition differs from the baseline table because of missing data.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Status Quo | Flavors Banned | Flavors and Menthol Banned
Number analyzed (Participants) | 74 | 74 | 75
proportion of participants | .34 [.22 to .48] | .35 [.23 to .50] | .42 [.28 to .57]
Statistical Analysis 1: Comparison: Status Quo vs Flavors Banned; Test type: Other; Odds Ratio (OR) = 1.08, 95% CI 2-sided [.47 to 2.49] — Adjusted for age, education, and lifetime use of tobacco
Statistical Analysis 2: Comparison: Status Quo vs Flavors and Menthol Banned; Test type: Other; Odds Ratio (OR) = 1.43, 95% CI 2-sided [.62 to 3.31] — Adjusted for age, education, and lifetime use of tobacco products

5. Secondary Outcome: Proportion of Participants Susceptible to Using Electronic Nicotine Delivery Device (ENDS) After Shopping in the StoreLab (Menthol-flavored)
Description: Self-report items: "Do you think you will try a vaping product flavored with menthol or mint soon?", "Do you think you will use a vaping product flavored with menthol or mint anytime in the next year?"; and "If one of your best friends offered you a vaping product flavored with menthol or mint, would you use it?". Responses to each item were made on a 1 (Definitely Not) to 10 (Definitely Yes) scale and the three items were summed. The total scale score was dichotomized: those who scored a '3' were recoded as '0' (not susceptible) and any scores greater than '3' were coded as '1' (susceptible). Proportion of susceptible participants was the outcome (number susceptible over the total number of participants within condition).
Time Frame: as for outcome 1
Population: The numbers of participants per condition differs from the baseline table because of missing data.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Status Quo | Flavors Banned | Flavors and Menthol Banned
Number analyzed (Participants) | 75 | 74 | 74
proportion of participants | .27 [.16 to .41] | .39 [.25 to .54] | .43 [.29 to .58]
Statistical Analysis 1: Comparison: Status Quo vs Flavors Banned; Test type: Other; Odds Ratio (OR) = 1.73, 95% CI 2-sided [.72 to 4.14] — Adjusted for age, education, and lifetime use of tobacco products
Statistical Analysis 2: Comparison: Status Quo vs Flavors and Menthol Banned; Test type: Other; Odds Ratio (OR) = 2.03, 95% CI 2-sided [.83 to 4.95] — Adjusted for age, education, and lifetime use of tobacco products

6. Secondary Outcome: Proportion of Participants Susceptible to Using Little Cigar/Cigarillos (LCC) After Shopping in the StoreLab (Non-flavored)
Description: Self-report items: "Do you think you will try an unflavored cigarillos/filtered cigar soon?", "Do you think you will use an unflavored cigarillos/filtered cigar anytime in the next year?"; and "If one of your best friends offered you an unflavored cigarillos/filtered cigar, would you use it?". Responses to each item were made on a 1 (Definitely Not) to 10 (Definitely Yes) scale and the three items were summed. The total scale score was dichotomized: those who scored a '3' were recoded as '0' (not susceptible) and any scores greater than '3' were coded as '1' (susceptible). Outcome is proportion of participants susceptible to using LCCs after shopping in the StoreLab (number susceptible over the total number of participants within condition).
Time Frame: as for outcome 1
Population: The numbers of participants per condition differs from the baseline table because of missing data.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Status Quo | Flavors Banned | Flavors and Menthol Banned
Number analyzed (Participants) | 74 | 73 | 74
proportion of participants | .09 [.04 to .19] | .10 [.05 to .21] | .17 [.09 to .31]
Statistical Analysis 1: Comparison: Status Quo vs Flavors Banned; Test type: Other; Odds Ratio (OR) = 1.13, 95% CI 2-sided [.40 to 3.18] — Adjusted for age, education, and lifetime tobacco use
Statistical Analysis 2: Comparison: Status Quo vs Flavors and Menthol Banned; Test type: Other; Odds Ratio (OR) = 2.04, 95% CI 2-sided [.73 to 5.71] — Adjusted for age, education, and lifetime tobacco use

7. Secondary Outcome: Proportion of Participants Susceptible to Using Little Cigar/Cigarillos (LCC) After Shopping in the StoreLab (Sweet-flavored)
Description: Self-report items: "Do you think you will try a cigarillos/filtered cigar flavored with fruit, candy, alcohol or some other sweet flavor soon?", "Do you think you will use a cigarillos/filtered cigar flavored with fruit, candy, alcohol or some other sweet flavor anytime in the next year?"; and "If one of your best friends offered you a cigarillos/filtered cigar flavored with fruit, candy, alcohol or some other sweet flavor would you use it?". Responses to each item were made on a 1 (Definitely Not) to 10 (Definitely Yes) scale and the three items were summed. The total scale score was dichotomized: those who scored a '3' were recoded as '0' (not susceptible) and any scores greater than '3' were coded as '1' (susceptible). Proportion of susceptible participants was the outcome (number susceptible over the total number of participants within condition).
Time Frame: as for outcome 1
Population: The numbers of participants per condition differs from the baseline table because of missing data.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Status Quo | Flavors Banned | Flavors and Menthol Banned
Number analyzed (Participants) | 74 | 73 | 75
proportion of participants | .10 [.05 to .19] | .16 [.08 to .28] | .25 [.14 to .39]
Statistical Analysis 1: Comparison: Status Quo vs Flavors Banned; Test type: Other; Odds Ratio (OR) = 1.77, 95% CI 2-sided [.66 to 4.75] — Adjusted for age, education, and lifetime tobacco use
Statistical Analysis 2: Comparison: Status Quo vs Flavors and Menthol Banned; Test type: Other; Odds Ratio (OR) = 3.06, 95% CI 2-sided [1.13 to 8.29] — Adjusted for age, education, and lifetime use of tobacco

8. Secondary Outcome: Proportion of Participants Susceptible to Using Little Cigar/Cigarillos (LCC) After Shopping in the StoreLab (Menthol-flavored)
Description: Self-report items: "Do you think you will try a cigarillos/filtered cigar flavored with menthol or mint soon?", "Do you think you will use a cigarillos/filtered cigar flavored with menthol or mint anytime in the next year?"; and "If one of your best friends offered you a cigarillos/filtered cigar flavored with menthol or mint would you use it?". Responses to each item were made on a 1 (Definitely Not) to 10 (Definitely Yes) scale and the three items were summed. The total scale score was dichotomized: those who scored a '3' were recoded as '0' (not susceptible) and any scores greater than '3' were coded as '1' (susceptible). Outcome is proportion of participants susceptible to using LCCs after shopping in the StoreLab (number of susceptible over number in condition).
Time Frame: as for outcome 1
Population: The numbers of participants per condition differs from the baseline table because of missing data.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Status Quo | Flavors Banned | Flavors and Menthol Banned
Number analyzed (Participants) | 74 | 74 | 75
proportion of participants | .10 [.05 to .20] | .13 [.07 to .25] | .21 [.11 to .35]
Statistical Analysis 1: Comparison: Status Quo vs Flavors Banned; Test type: Other; Odds Ratio (OR) = 1.38, 95% CI 2-sided [.51 to 3.70] — Adjusted for age, education, and lifetime tobacco use
Statistical Analysis 2: Comparison: Status Quo vs Flavors and Menthol Banned; Test type: Other; Odds Ratio (OR) = 2.32, 95% CI 2-sided [.85 to 6.31] — Adjusted for age, education, and lifetime tobacco use

9. Secondary Outcome: Proportion of Participants Susceptible to Using Smokeless Tobacco After Shopping in the StoreLab (Non-flavored)
Description: Self-report items: "Do you think you will try unflavored smokeless tobacco soon?", "Do you think you will use unflavored smokeless tobacco anytime in the next year?"; and "If one of your best friends offered you unflavored smokeless tobacco, would you use it?". Responses to each item were made on a 1 (Definitely Not) to 10 (Definitely Yes) scale and the three items were summed. The total scale score was dichotomized: those who scored a '3' were recoded as '0' (not susceptible) and any scores greater than '3' were coded as '1' (susceptible). Proportion of susceptible participants was the outcome (number susceptible over the total number of participants within condition).
Time Frame: as for outcome 1
Population: The numbers of participants per condition differs from the baseline table because of missing data.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Status Quo | Flavors Banned | Flavors and Menthol Banned
Number analyzed (Participants) | 75 | 68 | 73
proportion of participants | .06 [.03 to .15] | .07 [.03 to .17] | .12 [.06 to .24]
Statistical Analysis 1: Comparison: Status Quo vs Flavors Banned; Test type: Other; Odds Ratio (OR) = 1.11, 95% CI 2-sided [.29 to 4.26] — Adjusted for age, education, and lifetime tobacco use
Statistical Analysis 2: Comparison: Status Quo vs Flavors and Menthol Banned; Test type: Other; Odds Ratio (OR) = 2.00, 95% CI 2-sided [.57 to 7.06] — Adjusted for age, education, and lifetime tobacco use

10. Secondary Outcome: Proportion of Participants Susceptible to Using Smokeless Tobacco After Shopping in the StoreLab (Sweet-flavored)
Description: Self-report items: "Do you think you will try smokeless tobacco flavored with fruit soon?", "Do you think you will use smokeless tobacco flavored with fruit anytime in the next year?"; and "If one of your best friends offered you smokeless tobacco flavored with fruit, would you use it?". Responses to each item were made on a 1 (Definitely Not) to 10 (Definitely Yes) scale and the three items were summed. The total scale score was dichotomized: those who scored a '3' were recoded as '0' (not susceptible) and any scores greater than '3' were coded as '1' (susceptible). Proportion of susceptible participants was the outcome (number susceptible over the total number of participants within condition).
Time Frame: as for outcome 1
Population: The numbers of participants per condition differs from the baseline table because of missing data.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Status Quo | Flavors Banned | Flavors and Menthol Banned
Number analyzed (Participants) | 72 | 72 | 74
proportion of participants | .09 [.04 to .19] | .10 [.04 to .20] | .20 [.11 to .33]
Statistical Analysis 1: Comparison: Status Quo vs Flavors Banned; Test type: Other; Odds Ratio (OR) = 1.04, 95% CI 2-sided [.33 to 3.31] — Adjusted for age, education, and lifetime tobacco use
Statistical Analysis 2: Comparison: Status Quo vs Flavors and Menthol Banned; Test type: Other; Odds Ratio (OR) = 2.43, .95% CI 2-sided [.83 to 7.13] — Adjusted for age, education, and lifetime tobacco use

11. Secondary Outcome: Proportion of Participants Susceptible to Using Smokeless Tobacco After Shopping in the StoreLab (Menthol-flavored)
Description: Self-report items: "Do you think you will try smokeless tobacco flavored with menthol, mint, spearmint, or wintergreen soon?", "Do you think you will use smokeless tobacco flavored with menthol, mint, spearmint, or wintergreen anytime in the next year?"; and "If one of your best friends offered you smokeless tobacco flavored with menthol, mint, spearmint, or wintergreen, would you use it?". Responses to each item were made on a 1 (Definitely Not) to 10 (Definitely Yes) scale and the three items were summed. The total scale score was dichotomized: those who scored a '3' were recoded as '0' (not susceptible) and any scores greater than '3' were coded as '1' (susceptible). Proportion of susceptible participants was the outcome (number susceptible over the total number of participants within condition).
Time Frame: as for outcome 1
Population: The numbers of participants per condition differs from the baseline table because of missing data.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Status Quo | Flavors Banned | Flavors and Menthol Banned
Number analyzed (Participants) | 75 | 74 | 74
proportion of participants | .27 [.16 to .41] | .39 [.25 to .54] | .43 [.29 to .58]
Statistical Analysis 1: Comparison: Status Quo vs Flavors Banned; Test type: Other; Odds Ratio (OR) = 1.73, 95% CI 2-sided [.72 to 4.14] — Adjusted for age, education, and lifetime tobacco use
Statistical Analysis 2: Comparison: Status Quo vs Flavors and Menthol Banned; Test type: Other; Odds Ratio (OR) = 2.03, 95% CI 2-sided [.83 to 4.95] — Adjusted for age, education, and lifetime tobacco use

ADVERSE EVENTS:
Time Frame: Two hours
Arm/Group | Status Quo | Flavors Banned | Flavors and Menthol Banned
All-Cause Mortality (participants affected / at risk) | 0/89 | 0/91 | 0/87
Serious Adverse Events (participants affected / at risk) | 0/89 | 0/91 | 0/87
Other Adverse Events (participants affected / at risk) | 0/89 | 0/91 | 0/87

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-16): https://cdn.clinicaltrials.gov/large-docs/49/NCT04259749/Prot_SAP_000.pdf